CLINICAL TRIAL: NCT03385343
Title: Staging of Superficial Esophageal Adenocarcinoma (EAC) Using Volumetric Laser Endomicroscopy (VLE)
Brief Title: Staging of Superficial EAC Using VLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device company went out of business
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-002723
Record Dates: First submitted 2017-08-29; First posted 2017-12-28 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- VLE imaging of stage EAC (Experimental): All subjects will receive VLE imaging for staging EAC. Volumetric laser endomicroscopy (VLE) is an imaging platform that uses infrared light to generate cross-sectional views of the human esophagus with microscopic resolution.
  Interventions: Diagnostic Test: VLE imaging for staging EAC

INTERVENTIONS:
Diagnostic Test: VLE imaging for staging EAC — Volumetric Laser Endomicroscopy (VLE) imaging for staging Esophageal Adenocarcinoma (EAC)
  Other Names: NvisionVLE Imaging System

SUMMARY:
This study is being done to see if the NvisionVLE Imaging System can accurately determine the diagnostic performance of staging of T1 esophageal adenocarcinoma.

DETAILED DESCRIPTION:
Volumetric laser endomicroscopy (VLE) is an imaging platform that uses infrared light to generate cross-sectional views of the human esophagus with microscopic resolution. VLE has been used to detect dysplasia associated with Barrett's esophagus (BE) but its use in cancer staging has not been previously explored. The investigators propose that VLE can accurately and comprehensively stage T1 EAC.

VLE scans will be analyzed using an automated computer algorithm to measure degree of signal attenuation over areas demarcated for endoscopic mucosal resection (EMR). The signal attenuation cut-off established will be used to classify cancers as superficial versus deep. EMR specimens will be reviewed histopathologically for grade of tumor differentiation, depth of invasion, and presence or absence of lymphovascular invasion. Depth of tumor invasion will be measured and used to classify cancers as superficial versus deep.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* Patient undergoing an upper endoscopy with prior-biopsy confirmed Barrett's Esophagus.
* Ability to provide written, informed consent
* No significant esophagitis (LA grade <B, C, and D)

Exclusion Criteria:

* Patients who have achieved complete remission of intestinal metaplasia (CR-IM)
* Patients without visible Barrett's Esophagus at the time of study esophagogastroduodenoscopy (EGD)
* Patients for whom use of the NvisionVLE device would be in conflict with the instruction for use.
* Prior esophageal or gastric surgical resection
* Significant esophageal stricture requiring dilatation
* Patients who require anticoagulation for who biopsy would be contraindicated
* Patients who are known to be pregnant

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cadman L Leggett, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing clinical care through our institution's Barrett's esophagus unit.
Groups:
- Volumetric Laser Endomicroscopy: Patients with Barrett's esophagus and early esophageal adenocarcioma (T1) who were undergoing a clinically indicated endoscopic mucosal resection (EMR) were invited to participate in the study. EMR specimens were imaged (ex-vivo) using volumetric laser endomicroscopy (VLE).
Period: Overall Study
Arm/Group | Volumetric Laser Endomicroscopy
Started | 30
Completed | 22
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Volumetric Laser Endomicroscopy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 68.33 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose VLE Results Correlates With the Histology Results for T1 EAC Depth of Invasion
Description: A validated computer algorithm will be used to quantify the degree of signal attenuation in the T1 EAC endoscopic mucosal resection specimen database. Volumetric Laser Endo-microscopy (VLE) signal attenuation measurements will be correlated to depth of invasion as determined by histology.
Time Frame: 1 day
Population: Data was not collected
Arm/Group | Volumetric Laser Endomicroscopy
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Subjects Whose VLE Results Correlates With the Histology Results for Staging T1 EAC
Description: To validate the accuracy of VLE in staging T1 EAC compared to a histologic gold-standard.
Time Frame: 1 day
Population: Data was not collected
Arm/Group | VLE Imaging of Stage EAC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assessed due to ex-vivo nature of the study
Groups:
- VLE in Staging T1 EAC: The diagnostic performance of VLE in staging T1 EAC
Arm/Group | VLE in Staging T1 EAC
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03385343/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03385343/ICF_001.pdf